CLINICAL TRIAL: NCT03173365
Title: Half-Side Controlled Analysis of the Effect of Topical Brimonidine Tartrate on the Frequency and Severity of Hand-Foot Syndrome (HFS) in Cancer Patients Receiving Antineoplastic Agents (BRIMOCAN)
Brief Title: The Effect of Topical Brimonidine Tartrate on Hand-foot Syndrome (HFS) in Cancer Patients
Acronym: BRIMOCAN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: It is no longer practicable to complete the trial
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRIMOCAN
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Hand-foot Syndrome
Keywords: Hand-foot Syndrome; Brimonidine; Mirvaso; palmar-plantar erythrodysesthesia syndrome; Brimonidine Tartrate
MeSH Terms: conditions — Hand-Foot Syndrome | interventions — Brimonidine Tartrate

STUDY DESIGN:
Intervention Model Description: The respective palm to be treated will be randomly assessed and will be matched for handedness to include equal numbers of dominant and non-dominant treated palms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brimonidine Tartrate (Experimental): The respective palm to be treated with Brimonidine will be randomly assessed and will be matched for handedness to include equal numbers of dominant and non-dominant treated palms.
  Interventions: Drug: Brimonidine Tartrate

INTERVENTIONS:
Drug: Brimonidine Tartrate — 1 gram of Brimonidine 3 mg/g gel (Mirvaso®) in 24 hours on the randomized palm equal to a finger tip unit (FTU) of 0.5 gram , topical application under occlusion twice per day, every 12 hours.
  Other Names: Mirvaso

SUMMARY:
Comparative analysis of the severity of Hand-Foot-Syndrome (HFS) of palms treated with brimonidine tartrate gel or with standard care Urea 10% containing lotion in cancer patients receiving antineoplastic therapy to show a preventive effect of cutaneous brimonidine treatment on severity of HFS symptoms.

DETAILED DESCRIPTION:
Hand-foot syndrome (HFS) is an adverse event frequently associated with the use of classical chemotherapeutic agents such as capecitabine or pegylated liposomal doxorubicin, as well as targeted cancer drugs such as sorafenib or other tyrosine-kinase inhibitors. If the toxicity progresses edematous swelling, blistering and desquamation can lead to ulcerations of the palms and soles. Additionally, patients may be affected by nail-toxicities, such as discoloration, ridging, pitting up to complete onycholysis and pain. Today, cooling of hands and feet during infusion chemotherapy as well as preventive treatment with topical formulations containing urea 10% (e.g. Excipial U10 Lipolotion®) is considered as standard of care. Yet, these strategies are limited by intricateness, patient inconvenience and low efficacy. Hence, at this point the satisfactory treatment of HFS remains an unmet medical need, as until now, no effective therapy is available to prevent or reduce HFS symptoms during the cycle of chemotherapeutic treatment.

Recently, brimonidine 3 mg/g gel (Mirvaso®) has been approved as a topical treatment of facial erythema of rosacea in adult patients. Brimonidine is an effective agonist of α2-adrenoreceptors thereby, in analogy to skin cooling, leading to peripheral vasoconstriction.

Against this background, the following hypothesis was developed:

The topical application brimonidine 3 mg/g gel (Mirvaso®) may prevent or reduce the severity of HFS in cancer patients that receive respective antineoplastic agents.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients with solid tumors under antineoplastic therapy with capecitabine or pegylated liposomal doxorubicin.
* Patients with a life expectancy of at least 12 weeks.
* History of HFS (grades 2 to 3) in the course of the therapy
* Patients who are 18-65 years old.
* Regression of HFS to grade 1 or lower with a symmetrical grading on both hands (grade 0 or grade 1) prior to the next cycle of chemotherapy.
* not legally incapacitated
* Written informed consent from the trial subject has been obtained.
* Current treatment with capecitabine or pegylated liposomal doxorubicin

Exclusion Criteria:

* Persons with any kind of dependency on the investigator or employed by the sponsor or investigator.
* Persons held in an institution by legal or official order.
* Participation in other interventional trials
* Drug & substance abuse
* Use of central nervous depressants (e.g. alcohol, barbiturates, opiates, sedatives or anaesthetics)
* Patients taking alpha adrenergic agonists as medication.
* Pregnant women and nursing mothers
* Failure to use highly-effective contraceptive methods

The following contraceptive methods with a Pearl Index lower than 1% are regarded as highly effective:

* Oral hormonal contraception ('pill')
* Vaginal hormonal contraception (NuvaRing®)
* Contraceptive plaster
* Long-acting injectable contraceptives
* Implants that release progesterone (Implanon®)
* Tubal ligation (female sterilization)
* Intrauterine devices that release hormones (hormone spiral)
* Double barrier methods: This means that the following are not regarded as safe: condom plus spermicide, simple barrier methods (vaginal pessaries, condom, female condoms), copper spirals, the rhythm method, basal temperature method, and the withdrawal method (coitus interruptus).

  * History of inflammatory dermatosis of hands or feet (e.g. hand eczema)
  * Smoking
  * Severe or unstable or uncontrolled cardiovascular disease
  * Depression
  * cerebral or coronary insufficiency
  * Raynaud's phenomenon
  * orthostatic hypotension
  * thrombangiitis obliterans
  * Scleroderma
  * Sjögren's syndrome
  * renal or hepatic impairment
  * Known allergic sensitization against any of the substances applied in the study
  * Patients receiving monoamine oxidase (MAO) inhibitor therapy (for example selegiline or moclobemide) and patients on tricyclic (such as imipramine) or tetracyclic (such as maprotiline, mianserin or mirtazapin) antidepressants which affect noradrenergic transmission.
  * Patients receiving topical corticoids on hands or feet within 1 week prior to baseline measurement and during the entire study treatment period of up to six weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number and time of occurence of Palms with HFS severity grade 2 or 3 | weekly up to 6 weeks
  Palms with HFS severity of grade 2 or 3 during 2 cycles of chemotherapy or over 6 week period by means of the National Cancer Institute Common Terminology criteria for Adverse Events (NCI-CTCAE) v4.0 grading

SECONDARY OUTCOMES:
NCI-CTCAE v4.0 grading of HFS severity | weekly up to 6 weeks
  Severity of HFS after 2 cycles of chemotherapy or 6 weeks by means of the NCI-CTCAE v4.0 grading
Severity of nail toxicity | weekly up to 6 weeks
  Severity of nail toxicity after 2 cycles of chemotherapy or 6 weeks by means of the NCI-CTCAE v3.0 grading
modified ppPASI grading of HFS severity | weekly up to 6 weeks
  Severity of HFS after 2 cycles of chemotherapy or 6 weeks by means of a modified Palmoplantar Psoriasis Area Severity Index (ppPASI)
computer-assisted quantification of HFS severity | weekly up to 6 weeks
  Severity of HFS after 2 cycles of chemotherapy or 6 weeks by means of computer-assisted quantification
HFS associated pain (by VAS scale) | weekly up to 6 weeks
  Level of HFS-associated pain after 2 cycles of chemotherapy or 6 weeks by means of visual analogue scale (VAS)
Highest grade of HFS severity (NCI-CTCAE v4.0 grading) | weekly up to 6 weeks
  Highest grade of HFS severity reached until 2 cycle of chemotherapy or over 6 week period by means of the NCI-CTCAE v4.0 grading

CONTACTS AND LOCATIONS:
Overall Officials: Peter Arne Gerber, PD Dr. med., Principal Investigator — Heinrich-Heine University, Duesseldorf
Locations (1):
- Universitätsklinikum Düsseldorf, Klinik für Dermatologie, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No